CLINICAL TRIAL: NCT05096910
Title: COSMOSS Study, Comparison Of Suture Materials on Sectio Scars. A Multicenter Prospective Randomized Controlled Study
Brief Title: Comparison Of Suture Materials on Sectio Scars (COSMOSS)
Acronym: COSMOSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uludag University (Other)
Collaborators: Medicana Bursa Hospital (Other); UMI Health Center (Unknown); Ceylan Hospital (Unknown)
Responsible Party: Principal Investigator, GÜRKAN UNCU,PROF. MD, M.D, Professor, Uludag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10840098-772.02-E.43598
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Uterine Scar
Keywords: cesarean section; isthmocele; uterine scar; suture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monofilament Suture Group (Active Comparator): Monofilament sutures will be used for uterine closure.
  Interventions: Procedure: Uterine Closure with monofilament or polyfilament suture materials
- Polyfilament Suture Group (Active Comparator): Polyfilament sutures will be used for uterine closure.
  Interventions: Procedure: Uterine Closure with monofilament or polyfilament suture materials

INTERVENTIONS:
Procedure: Uterine Closure with monofilament or polyfilament suture materials — Postoperative 6th-month isthmocele rates

SUMMARY:
This multicenter prospective randomized controlled trial aims to investigate the ishtmocele rates after c-section delivery depending on using different suture materials for the uterine closure.

DETAILED DESCRIPTION:
The study involves 5 health centers (two universities, three private hospitals). Patients who will undergo their first cesarean section because of any etiology (except emergent cases) will be included in the study. Operation Nurse will randomize the patients into two groups depending on the monofilament or poly filament suture material. Patients will be checked by transvaginal ultrasound on a postoperative day one, postoperative first month, and postoperative sixth month. As the primary result, the istmocele rates will be compared between the study groups.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 yrs women
* Primary elective cesarean section
* First delivery
* Without any systemic diseases

Exclusion Criteria:

* emergent delivery
* previous c-section history
* congenital uterine abnormality

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Isthmocele Rate | 6 months
  diagnosis of isthmocele during 6th month ultrasound check.

CONTACTS AND LOCATIONS:
Overall Officials: Gurkan Uncu, Prof., Study Director — Bursa Uludag University Faculty of Medicine
Locations (1):
- Uludag University Scholl of medicine, Bursa, Turkey/bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided